CLINICAL TRIAL: NCT00925067
Title: Effects of Lightweight Meshes in Laparoscopic Inguinal Hernia Repair on Quality of Life and Male Fertility Aspects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Fund for Scientific Research, Flanders, Belgium (Other); Agentschap voor Innovatie door Wetenschap en Technologie (Other)
Responsible Party: Marc Miserez, University Hospitals Leuven
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: G.0457.04N
Record Dates: First submitted 2009-06-18; First posted 2009-06-19 (Estimated); Last update posted 2009-06-19 (Estimated); Status verified 2009-06

CONDITIONS: Inguinal Hernia
Keywords: Inguinal hernia; Laparoscopic repair; Prostheses; Male fertility
MeSH Terms: conditions — Hernia, Inguinal | interventions — Laparoscopy; tetraethylpyrazine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- lightweight TiMesh (Experimental)
  Interventions: Procedure: laparoscopic (TEP) inguinal hernia repair; Device: lightweight TiMesh
- lightweight VyproII (Experimental)
  Interventions: Procedure: laparoscopic (TEP) inguinal hernia repair; Device: lightweight VyproII
- Heavyweight Marlex (Experimental)
  Interventions: Procedure: laparoscopic (TEP) inguinal hernia repair; Device: Heavyweight Marlex

INTERVENTIONS:
Procedure: laparoscopic (TEP) inguinal hernia repair — laparoscopic inguinal hernia repair with a standard heavyweight Marlex (control group) prosthesis or new generation lightweight VyproII and TiMesh prostheses (study group)
Device: lightweight TiMesh
  Arms: lightweight TiMesh
Device: lightweight VyproII
  Arms: lightweight VyproII
Device: Heavyweight Marlex
  Arms: Heavyweight Marlex

SUMMARY:
A randomized, prospective clinical trial analyzing whether the use of lightweight prostheses during laparoscopic inguinal hernia repair of male patients could have a beneficial effect on postoperative discomfort, chronic pain development, recurrence and male fertility aspects.

ELIGIBILITY:
Inclusion Criteria:

* Primary, unilateral or bilateral, inguinal hernia patients
* Informed consent

Exclusion Criteria:

* Sterilized patients

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2003-04; Primary Completion 2007-10 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Male fertility aspects | 12 months

SECONDARY OUTCOMES:
Quality of life, pain development, recurrence | 1, 3, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Marc Miserez, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Vlaams-Brabant, Belgium

REFERENCES:
- [Derived] Peeters E, Spiessens C, Oyen R, De Wever L, Vanderschueren D, Penninckx F, Miserez M. Laparoscopic inguinal hernia repair in men with lightweight meshes may significantly impair sperm motility: a randomized controlled trial. Ann Surg. 2010 Aug;252(2):240-6. doi: 10.1097/SLA.0b013e3181e8fac5. PMID 20622657